CLINICAL TRIAL: NCT05436834
Title: An Open-Label, Phase 3 Study to Evaluate the Safety and Immunogenicity of mRNA Vaccines for SARS-CoV-2 Variants in Participants Aged 6 Months to < 6 Years
Brief Title: A Study to Evaluate the Safety and Immunogenicity of the mRNA COVID-19 Vaccines in Healthy Children Between 6 Months to Less Than 6 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: mRNA-1273-P306
Record Dates: First submitted 2022-06-27; First posted 2022-06-29 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: SARS-CoV-2
Keywords: Coronavirus disease 2019; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — mRNA-1273.214 COVID-19 vaccine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- mRNA-1273.214 (Part 1) (Experimental): Participants who have not been previously vaccinated against SARS-CoV-2, will receive 2 intramuscular (IM) injections of mRNA-1273.214 vaccine on Day 1 and Day 29.
  Interventions: Biological: mRNA-1273.214
- mRNA-1273.214 (Part 2) (Experimental): Participants who have previously been vaccinated with a mRNA-1273 primary series, will receive a single IM BD of mRNA-1273.214 vaccine at least 4 months after completion of the mRNA-1273 primary series.
  Interventions: Biological: mRNA-1273.214
- mRNA-1273.815 (Part 3) (Experimental): Participants who have previously been vaccinated with an authorized/approved COVID-19 vaccine, will receive a single IM BD of mRNA-1273.815 vaccine on BD Day 1, at least 4 months after the last dose of a COVID-19 vaccine.
  Interventions: Biological: mRNA-1273.815
- mRNA-1273.815 (Part 4) (Experimental): Participants in Part 4 Cohort A will receive a single IM injection of mRNA-1273.815 vaccine on Day 1. Participants in Part 4 Cohort B will receive IM injections of mRNA-1273.815 vaccine on Day 1 and Day 29.
  Interventions: Biological: mRNA-1273.815

INTERVENTIONS:
Biological: mRNA-1273.214 — Sterile liquid for injection
  Arms: mRNA-1273.214 (Part 1); mRNA-1273.214 (Part 2)
Biological: mRNA-1273.815 — Sterile liquid for injection
  Arms: mRNA-1273.815 (Part 3); mRNA-1273.815 (Part 4)

SUMMARY:
This study will evaluate the safety and immunogenicity of the mRNA-1273.214 vaccine for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) variant of concerns (VOCs) in participants aged 6 months to <6 years, when administered as a primary series in SARS-CoV-2 vaccine-naïve participants (Part 1) and a single booster dose (BD) given to participants who previously received 2 doses of the mRNA-1273 vaccine as a primary series (Part 2); and will evaluate the safety and immunogenicity of the mRNA-1273.815 vaccine, when administered as a BD in participants aged 6 months to <6 years (Part 3) and when administered to SARS-CoV-2 vaccine-naïve participants aged 2 years to <5 years of age (Part 4).

DETAILED DESCRIPTION:
Part 1 will enroll participants aged 6 months to <6 years who have not been previously vaccinated against SARS-CoV-2. Participants will receive 2 doses of the mRNA-1273.214 vaccine.

Part 2 will enroll participants aged 6 months to <6 years who have previously been vaccinated with a mRNA-1273 primary series in Study mRNA-1273-P204 (NCT04796896). Participants will receive a single BD of the mRNA-1273.214 vaccine, at least 4 months after completion of the mRNA-1273 primary series.

Part 3 will enroll participants aged 6 months to <6 years who have previously been vaccinated with an authorized/approved COVID-19 vaccine. Participants will receive a BD of the mRNA-1273.815 vaccine at least 4 months after the last receipt of a COVID-19 vaccine.

Part 4 will evaluate mRNA-1273.815 vaccine administered as a single dose to SARS-CoV-2 vaccine-naïve participants aged 2 years to <5 years of age enrolled in Cohort A (Part 4A), compared to 2 doses given to SARS-CoV-2 vaccine-naïve participants aged 6 months to <2 years enrolled in Cohort B (Part 4B).

ELIGIBILITY:
Inclusion Criteria:

* The participant is 6 months to <6 years for Parts 1, 2, and 3; 2 years to <5 years for Part 4A; and 6 months to <2 years for Part 4B at the time of consent (Screening Visit). Note: for Part 1, participant must be at least 6 months old and must not have reached 6 years of age at the time of administration of first dose. For Part 4B, the participant must be at least 6 months old and must not have reached 2 years of age at the time of administration of first dose.
* If the participant has a chronic disease (that is, asthma, diabetes mellitus, cystic fibrosis, human immunodeficiency virus [HIV] infection), the disease should be stable, per investigator assessment, so that the participant can be considered eligible for inclusion. Stable diseases are those which have had no change in their status or in the medications required to control them in the 6 months prior to Screening Visit. Note: a change in medication for dose optimization (that is, insulin dose changes, adjustments for age-related weight gain), change within class of medication, or reduction in dose are not considered signs of instability.
* In the investigator's opinion, the parent(s)/legally authorized representative(s) (LAR[s]) understand and are willing and physically able to comply with protocol-mandated follow-up, including all procedures and provide written informed consent.
* The participant is 2 years or older and has a body mass index (BMI) at or above the second percentile according to World Health Organization (WHO) Child Growth Standards at the Screening Visit.

OR

* The participant is less than 2 years of age and the participant's height and weight are both at or above the second percentile according to WHO Child Growth Standards at the Screening Visit.

Special inclusion criteria for participants aged 6 months to < 12 months:

* The participant was born at full-term (≥ 37 weeks gestation) with a minimum birth weight of 2.5 kilograms (kg).

Inclusion criteria for Part 2:

* The participant must have received 2 doses of mRNA-1273, approximately 28 to 35 days apart, as 25-μg primary series, and second dose was given at least 4 months prior to enrollment.

Inclusion criteria for Part 3 only:

- The participant must have received an age-appropriate immunization series of an authorized/approved COVID-19 vaccine, with the last dose given at least 4 months prior to enrolment (Previous vaccines NOT allowed are: XBB.1.5-containing formulation).

Exclusion Criteria:

* Has a known history of SARS-CoV-2 infection (that is, reported AE of COVID-19 or asymptomatic SARS-CoV-2 infection during Study mRNA-1273-P204 at the time of rollover into mRNA-1273-P306 or during Part 1 at the time of rollover into Part 3) in the 90 days prior to dosing in this study.
* Is acutely ill or febrile 24 hours prior to or at the Screening Visit. Fever is defined as a body temperature ≥ 38.0°Celsius (C)/≥ 100.4°Fahrenheit (F). Participants who meet this criterion may have visits rescheduled within the relevant study visit windows. Afebrile participants with minor illnesses can be enrolled at the discretion of the investigator.
* For Parts 1 and 4, participant has previously been administered an investigational or approved CoV (that is, SARS-CoV-2, SARS-CoV, Middle East respiratory syndrome coronavirus [MERS-CoV]) vaccine. For Part 2, participant who received any approved/investigational CoV vaccine are ineligible to participate except for those who received mRNA-1273 (prototype) vaccine.
* Has undergone treatment with investigational or approved agents for prophylaxis against COVID-19 (including receipt of SARS-CoV-2 monoclonal antibodies for prophylaxis or treatment) within 90 days prior to enrollment.
* Has a known hypersensitivity to a component of the vaccine or its excipients. Hypersensitivity includes, but is not limited to, anaphylaxis or immediate allergic reaction of any severity to a previous dose of an mRNA COVID-19 vaccine or any of its components (including polyethylene glycol [PEG] or immediate allergic reaction of any severity to polysorbate).
* Has a medical or psychiatric condition that, according to the investigator's judgment, may pose additional risk as a result of participation, interfere with safety assessments, or interfere with interpretation of results.
* Has a history of diagnosis or condition that, in the judgment of the investigator, may affect study endpoint assessment or compromise participant safety, specifically the following:

  * Congenital or acquired immunodeficiency, other than well-controlled HIV infection.
  * Chronic hepatitis or suspected active hepatitis
  * A bleeding disorder that is considered a contraindication to IM injection or phlebotomy
  * Dermatologic conditions that could affect local solicited AR assessments
  * Any prior diagnosis of malignancy (excluding nonmelanoma skin cancer)
* Has received the following:

  * Any routine vaccination with inactivated or live vaccine(s) within 14 days prior to study vaccination or plans to receive such a vaccine through 14 days following study vaccination.

Note: This excludes influenza vaccine that may be given anytime, but ideally at least 7 days before study dose. If a participant receives an influenza vaccine, this should be captured within the concomitant medication electronic case report form (eCRF).

* Systemic immunosuppressants or immune-modifying drugs for >14 days in total within 6 months prior to the day of enrollment (for corticosteroids, ≥1 milligrams (mg)/kg/day or ≥ 10 mg/day prednisone equivalent, if participant weighs >10 kg). Participants may have visits rescheduled for enrollment if they no longer meet this criterion within the Screening Visit window. Inhaled, nasal, and topical steroids, and palivizumab are allowed.
* Intravenous (IV) or subcutaneous (SC) blood products (red cells, platelets, immunoglobulins) within 3 months prior to enrollment.

Note: Other inclusion and exclusion criteria may apply.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1807 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Solicited Local and Systemic Adverse Reactions (ARs) | Up to Day 8 (7 days post-vaccination)
Number of Participants with Unsolicited Adverse Events (AEs) | Up to Day 29 (28 days after each injection)
Number of Participants with Medically-Attended AEs (MAAEs) | Up to Day 394 (12 months after last dose)
Number of Participants with Serious AEs (SAEs) | Up to Day 394 (12 months after last dose)
Number of Participants with Adverse Events of Special Interest (AESI) | Up to Day 394 (12 months after last dose)
Number of Participants with AEs Leading to Withdrawal | Up to Day 394 (12 months after last dose)
Geometric Mean (GM) of the Serum Antibody (Ab) Level against Omicron BA.1 and Ancestral SARS-CoV-2 after mRNA-1273.214 Administration at Day 57 | Day 57
GM of the Serum Ab Level against Omicron BA.1 and Ancestral SARS-CoV-2 after mRNA-1273.214 Administration at Day 29 | Day 29
Seroresponse Rate (SRR) against Omicron BA.1 and Ancestral SARS-CoV-2 after mRNA-1273.214 Administration | Day 29
GM of the Serum Ab Level against Omicron XBB.1.5 after mRNA-1273.815 Administration | Up to Day 57

SECONDARY OUTCOMES:
SRR against Omicron BA.1 and Ancestral SARS-CoV-2 after mRNA-1273.214 Administration Regardless of prior SARS-CoV-2 Infection | Day 57
GM of the Serum Ab Level against Omicron XBB.1.5 after mRNA-1273.815 Administration Regardless of prior SARS-CoV-2 Infection | Up to Day 57
SRR against Omicron XBB.1.5 after mRNA-1273.815 Administration Regardless of prior SARS-CoV-2 Infection | Up to Day 57

CONTACTS AND LOCATIONS:
Locations (74):
- United States (48):
  - Trinity Clinical Research, LLC, Bessemer, Alabama
  - Velcocity Clinical Research, Banning, California
  - Sera Collection Research Services, Montebello, California
  - Center For Clinical Trials LLC -Paramount, Paramount, California
  - University of Colorado, Aurora, Colorado
  - Meridian Clinical Research, Washington D.C., District of Columbia
  - Prohealth Research Center, Doral, Florida
  - University of Florida Jacksonville, Jacksonville, Florida
  - Kissimmee Clinical Research, Kissimmee, Florida
  - Med-Care Research, Miami, Florida
  - University of South Florida, Tampa, Florida
  - IResearch, Decatur, Georgia
  - Meridian Clinical Research, Macon, Georgia
  - Velcocity Clinical Research, Meridian, Idaho
  - Lurie Childrens Hospital, Chicago, Illinois
  - Meridian Clinical Research, Overland Park, Kansas
  - Michael W. Simon MD, PSC, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Velocity Clinical Research - Lafayette - PPDS, Lafayette, Louisiana
  - MedPharmics, Metairie, Louisiana
  - Velocity Clinical Research - Covington - PPDS, Metairie, Louisiana
  - Clinical Research Institute, Minneapolis, Minnesota
  - University of Missouri Health Care, Columbia, Missouri
  - Meridian Clinical Research, Hastings, Nebraska
  - Meridian Clinical Research, Lincoln, Nebraska
  - Be Well Clinical Studies, LLC - Lincoln - ERN - PPDS, Lincoln, Nebraska
  - Quality Clinical Research, Omaha, Nebraska
  - Velocity Clinical Research, Albuquerque, New Mexico
  - Meridian Clinical Research, Binghamton, New York
  - WellNow Urgent Care Clinical Research, East Amherst, New York
  - Child Healthcare Associates - East Syracuse, East Syracuse, New York
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Velcocity Clinical Research, East Greenwich, Rhode Island
  - Coastal Pediatric Associates, Charleston, South Carolina
  - Meridian Clinical Research, Charleston, South Carolina
  - MUSC, Charleston, South Carolina
  - Le Bonheur Childrens Hospital, Memphis, Tennessee
  - Velocity Clinical Research Austin, Austin, Texas
  - REX Clinical Trials, LLC Beaumont, Beaumont, Texas
  - Velcocity Clinical Research, Cedar Park, Texas
  - BRCR Global Texas, Edinburg, Texas
  - Village Health Partners - Frisco Medical Village, Frisco, Texas
  - Ventavia Research Group, Houston, Texas
  - Cyfair Clinical Reseach Center, Houston, Texas
  - Texas Center for Drug Development, Houston, Texas
  - Victoria Clinical Research Group, Victoria, Texas
  - PI Coor Clinical Research LLC, Burke, Virginia
  - Clinical Research Partners, Richmond, Virginia
- Argentina (4):
  - AES - AS - Glenny Corp. S.A. Buenos Aires, CABA, Buenos Aires F.D.
  - Hospital Militar Central Cirujano Mayor Dr. Cosme Argerich, Buenos Aires, Ciudad Autónoma de BuenosAires
  - AES - AS - Clinica Mayo de Urgencias, San Miguel de Tucumán, Tucumán Province
  - Consultorios Médicos Dr. Doreski - PPDS, Buenos Aires
- Centro de Estudios Clinicos e Investigaciones Medicas (CECIM), Santiago, Santiago Metropolitan, Chile
- Colombia (8):
  - AES - AS - Centro de Investigación Clínica CIC S.A.S (CECIC) Medellín, Medellín, Antioquia
  - Clínica de Costa S.A.S, Barranquilla, Atlántico
  - AES- AS- Solano & Terront Servicios Médicos LTDA (UNIENDO) Bogotá, Bogotá, Bogota D.C.
  - Centro de Atencion e Investigacion Medica S.A.S. - CAIMED Aguazul, Aguazul, Casanare Department
  - Centro de Atencion e Investigacion Medica S.A - Yopal - CAIMED, Yopal, Casanare Department
  - Policlínico Social del Norte, Bogotá, Cundinamarca
  - Clínica de la Costa S.A.S- Sede Cartagena, Cartagena, Departamento de Bolívar
  - Centro de Atención e Investigación Médica S.A.S.- CAIMED - S.A.S. Sede Acacias, Acacías, Meta Department
- Dominican Republic (5):
  - Caimed Dominicana S.A.S - CAIMED - PPDS, Santo Domingo, Distrito NacionalSanto Domingo
  - Registrum- La Altagracia, Salvaleón de Higüey, La Altagracia Province
  - Hospital Materno Infantil San Lorenzo de Los Mina, Santo Domingo Este, Santo Domingo Province
  - Hospital General Regional Dr. Marcelino Velez Santana, Santo Domingo Iesta, Santo Domingo Province
  - Unidad de Vacunas e Investigación Instituto Dermatologico Dominicano y Cirugía de Piel Dr. Huberto B, Santo Domingo
- Panama (7):
  - CAENSA Clinical Trial, Panama City
  - Centro De Vacunacion Internacional, S.A. - David - Cevaxin - PPDS, Panama City
  - CEVAXIN 24 de diciembre - PPDS, Panama City
  - CEVAXIN Avenida México - PPDS, Panama City
  - CEVAXIN Chorrera - PPDS, Panama City
  - Curaex Clinical Trial, Panama City
  - Instituto de Investigaciones Científicas y Servicios de Alta Tecnología Asociación de Interés Panama, Panama City
- Caribbean Medical Research Center, San Juan, Puerto Rico

REFERENCES:
- [Derived] Dixit A, Bennett R, Ali K, Griffin C, Clifford RA, Turner M, Poston R, Hautzinger K, Yeakey A, Girard B, Zhou W, Deng W, Zhou H, Schnyder Ghamloush S, Kuter BJ, Slobod K, Miller JM, Priddy F, Das R; ROVER Study Investigators. Interim safety and immunogenicity of COVID-19 omicron BA.1 variant-containing vaccine in children in the USA: an open-label non-randomised phase 3 trial. Lancet Infect Dis. 2024 Jul;24(7):687-697. doi: 10.1016/S1473-3099(24)00101-4. Epub 2024 Mar 19. PMID 38518789